CLINICAL TRIAL: NCT04370197
Title: Impact of th Covid-19 Epidemic on Acute Stroke Management
Brief Title: Covid-19 Epidemic on Acute Stroke Management
Acronym: Stroke-Covid19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7826
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Stroke, Acute
Keywords: STROKE , Acute; Covid-19; SARS-COV-2; Mechanical thrombectomy; Thrombolysis
MeSH Terms: conditions — Stroke; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Covid-19 pandemic is a pandemic of an emerging infectious disease, coronavirus 2019 (Covid-19), caused by the coronavirus SARS-CoV-2. It appears in November 2019 in the city of Wuhan, China, and spreads worldwide from February 2020. The first cases of infection in France were confirmed on 24 January 2020. As of April 14, 103,573 cases of infection were confirmed, 32,292 hospitalized cases, including 6,730 in intensive care, with 15,729 deaths recorded1. The most affected regions are Ile de France and the Grand Est (in particular the Haut-Rhin department). Containment of the entire French population was introduced on 17 March, with the aim of reducing the spread of the virus and relieving the burden on the health system, particularly the intensive care units.

This unprecedented health crisis, as well as the social containment measures in themselves, has repercussions on other acute medical pthologies, not directly related to the viral infection. It appears that the number of patients treated for acute stroke has suddenly declined since the beginning of the epidemic.

However, it is not clear whether it is the incidence of stroke that has declined or simply the proportion of patients presenting within the time frame that allows for treatment in the acute phase (by thrombolysis or thrombectomy).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Stroke Patients
* Patient who agreed to participate in this study

Exclusion Criteria:

- Refusal to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Study of the effect of pandemic covid-19 on the management of stroke patients | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Neuroradiologie Interventionnelle, Strasbourg, France